CLINICAL TRIAL: NCT00229086
Title: Long Term Follow-up European Gatekeeper Study 005
Brief Title: Gatekeeper European 005
Status: Terminated | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Other Study IDs: MGU-004
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

INTERVENTIONS:
Device: Gatekeeper Reflux Repari System (Device)

SUMMARY:
Evaluation of the Gatekeeper System in the treatment of patients with Gastroesophageal Reflux Disease (GERD) who already have been treated under study protocols Endo 2000-03 and Endo 2000-04

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have been part of the Endo 2000-03 or Endo 2000-04 clinical study
* Subjects who have been informed of the nature of the long-term follow-up study and have agreed to its participation and provided Informed Consent

Exclusion Criteria:

* Underwent another endoscopic or surgical treatment for GERD (except re-intervention with Gatekeeper)
* Developed other medical illness that may cause the subject to be non-compliant
* Extensive Barrett's Esophagus (>2 cm)
* Unable or unwilling to cooperate with the study procedures

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 55

CONTACTS AND LOCATIONS:
Overall Officials: Medtronic GU Investigator, Principal Investigator — MedtronicNeuro
Locations (2):
- Contact Medtronic for specific site information, Minneapolis, Minnesota, United States
- Contact Medtronic for specific location, Tolochenaz, Switzerland